CLINICAL TRIAL: NCT01062971
Title: Comparative Clinical Study of The Safety And Efficacy of A New Fixed-Combination of Timolol-Brimonidine-Dorzolamide In Patients With Open Angle Glaucoma Or Ocular Hypertension
Brief Title: Clinical Study of A Fixed Combination of Timolol-Brimonidine-Dorzolamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Leopoldo Baiza-Duran, Laboratorios Sophia S.A de C.V.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPHIA-PRO-122
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; Ocular hypertension; POAG; Treatment
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): IOP Dorzolamide-Timolol-Brimonidine group
  Interventions: Drug: dorzolamide-timolol-brimonidine
- B (Active Comparator): IOP dorzolamide-timolol group
  Interventions: Drug: dorzolamide-timolol-brimonidine

INTERVENTIONS:
Drug: dorzolamide-timolol-brimonidine — Patients will be randomly divided into 2 groups, one of them treated with a new formulation of 0.5% timolol-0.2% brimonidine-2% dorzolamide in fixed combination (Krytantek Ofteno®, Laboratorios Sophia, Mexico) and the other one treated with 0.5% timolol-2% dorzolamide fixed combination (Cosopt®, MSD Laboratories, USA). Patients will received 1 drop twice a day of either formulations.
  Other Names: Krytantek Ofteno; Cosopt

SUMMARY:
To compare intraocular pressure lowering effectiveness of a new fixed combination drug.

DETAILED DESCRIPTION:
This is a multicentric, double blind and prospective clinical study. We will include patients with confirmed diagnosis of primary open-angle glaucoma and/or ocular hypertension, with intraocular pressure (IOP) ranging between 21 and 31 mm Hg. Patients will be randomly divided into 2 groups, one of them treated with a new formulation of 0.5% timolol-0.2% brimonidine-2% dorzolamide in fixed combination (Krytantek Ofteno®, Laboratorios Sophia, Mexico) and the other one treated with 0.5% timolol-2% dorzolamide fixed combination (Cosopt®, MSD Laboratories, USA). Patients will receive 1 drop twice a day of either formulations and were examined at days 2, 7, 15, 30, 60, and 90 after initiation of treatment. The primary objective is to compare the efficacy of both formulations, estimated as a decrease in IOP. A Goldmann applanation tonometer will be used for IOP determination.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of either sex and any race with open-angle glaucoma or ocular hypertension;
* Visual acuity of 20/40 to 20/80 or better (Snellen equivalent).

Exclusion Criteria:

* Clinically relevant ophthalmic or systemic conditions may be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo M Baiza-Duran, MD, Study Director — Clinical Research Department. Laboratorios Sophia S.A de C.V.
Locations (1):
- Instituto de la Visión. Hospital Universitario La Carlota. Universidad de Montemorelos, Montemorelos, Nuevo León, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- A (Triple Therapy): Dorzolamide-Timolol-Brimonidine group
- B (Doble Therapy): dorzolamide-timolol group
Period: Overall Study
Arm/Group | A (Triple Therapy) | B (Doble Therapy)
Started | 60 | 63
Completed | 56 | 56
Not Completed | 4 | 7
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | A (Triple Therapy) | B (Doble Therapy) | Total
Number analyzed (Participants) | 56 | 56 | 112
Number analyzed (eyes) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.2) | 59.8 (12.5) | 60.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: subjects]
  european | 6 | 4 | 10
  african | 0 | 1 | 1
  hispanic | 48 | 50 | 98
  asian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Mexico | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: the intraocular pressure was measured by the Goldman tonometer and reported in millimeters of mercury.
Time Frame: basal (day 1 ) and final (day 60)
Population: the analysis of the groups was by protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A (Triple Therapy) | B (Doble Therapy)
Number analyzed (Participants) | 56 | 56
mmHg
  baseline | 24.1 (2.6) | 23.6 (2.2)
  Final | 13.9 (2.9) | 16.9 (3.4)
Statistical Analysis 1: Comparison: A (Triple Therapy) vs B (Doble Therapy); Test type: Non-Inferiority — Noninferiority was determined if the treatments did not show differences greater than 20%; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Adverse Events
Description: the numbers of adverse events were quantified by group of studies, the presence of each event was taken as a event.
Time Frame: basal (day 1 ) and security call (day 75)
Population: the analysis of the study groups was done by protocol
Measure: Number; unit: events
Arm/Group | A (Triple Therapy) | B (Doble Therapy)
Number analyzed (Participants) | 56 | 56
events | 2 | 6
Statistical Analysis 1: Comparison: A (Triple Therapy) vs B (Doble Therapy); Test type: Non-Inferiority — Noninferiority was determined if the treatments did not show differences greater than 20%; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: the evaluation of the adverse events was made during the 60 days of treatment and in a safety call at 15 days after the end of the clinical stage
Arm/Group | A (Triple Therapy) | B (Doble Therapy)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 2/56 | 6/56
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (Triple Therapy) (N=56) | B (Doble Therapy) (N=56)
ocular pain (Eye disorders) | 1 (1) | 3 (3)
ocular burning (Eye disorders) | 1 (1) | 2 (2)
chemosis (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
only the sponsor can publish the results of the authorization, if the IP wishes to report or discuss the results, it must request the sponsor a signed agreement.